CLINICAL TRIAL: NCT02670421
Title: Stress Management Intervention in Women's Heart Clinic, Heart SMART Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Anjali Bhagra, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-000081
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face to face Heart SMART program (Active Comparator): Stress management program presented in a face to face meeting of 90-100 minutes with daily printed program instructions to follow over the next 12 weeks, accompanied by reading from a book entitled The Mayo Clinic Guide to Stress Free Living.
  Interventions: Behavioral: Face to Face Heart SMART Program; Behavioral: Mayo Clinic Guide to Stress Free Living
- Online Heart SMART program (Active Comparator): Stress management program in the form of 10- minute videos completed weekly by participant on-line for 12 weeks, accompanied by reading from a book entitled The Mayo Clinic Guide to Stress Free Living.
  Interventions: Behavioral: On-line Heart SMART Program; Behavioral: Mayo Clinic Guide to Stress Free Living

INTERVENTIONS:
Behavioral: Face to Face Heart SMART Program — The Heart SMART stress management program survey consists of Perceived Stress Scale (PSS), Brief Resilience Scale (BRS), Patient Health Questionnaire (PHQ - 9) and Generalized Anxiety Disorder (GAD - 7), followed by email communication every three weeks.
  Arms: Face to face Heart SMART program
Behavioral: On-line Heart SMART Program — The Heart SMART stress management program survey consists of PSS (Perceived Stress Scale), BRS (Brief Resilience Scale), PHQ-9 (Patient Health Questionnaire) and GAD-7 (Generalized Anxiety Disorder) taken on-line in twelve, 10 minutes sessions.
  Arms: Online Heart SMART program
Behavioral: Mayo Clinic Guide to Stress Free Living — All subjects will be provided with a copy of the book entitled Mayo Clinic Guide to Stress Free Living and encouraged to read it over the twelve week study period.

SUMMARY:
Will the intervention (Heart SMART program) be feasible in moderate or high stress patients, who are referred to the Women's Heart and Preventive Cardiology clinics at Mayo Clinic?

DETAILED DESCRIPTION:
The Heart SMART Program is designed to offer a practical and efficacious stress management and resiliency intervention. It involves making participants aware of practices to enhance present moment awareness and engagement. It teaches learners to train their attention, and refine interpretation; utilizing principles of gratitude, compassion, acceptance, higher meaning and forgiveness. Participants will choose to use one of two delivery methods (either the face to face method or the on-line method) of the Heart SMART program.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 25-75 years.
2. Able to speak English and complete questionnaire.
3. Self-reported Stress Scale 6 - 10 (visual analog scale of 1 to 10 with 1 being lowest stress and 10 being highest stress)
4. Women in face to face session will have to be able to attend the SMART session.
5. Women in the online group will be required to have the ability to use internet to access the online training material.

Exclusion Criteria:

1. Self-reported Stress Index <6
2. Pregnant women will be excluded from participation in the study. Pregnancy test is not required because the intervention in this study poses no risk
3. Unable to give written consent
4. Inability or refusal to cooperate with study procedures

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in Heart SMART Program survey score | Baseline and 12 weeks

SECONDARY OUTCOMES:
Participant's adherence survey score to Heart SMART program | 16, 20 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Bhagra, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No